CLINICAL TRIAL: NCT01644188
Title: A Randomized, Double-Blind, Parallel Group Study to Evaluate the Efficacy and Safety of SAR236553/REGN727 Versus Ezetimibe in High Cardiovascular Risk Patients With Hypercholesterolemia Not Adequately Controlled With Their Statin Therapy
Brief Title: Efficacy and Safety of Alirocumab (SAR236553/REGN727) Versus Ezetimibe on Top of Statin in High Cardiovascular Risk Patients With Hypercholesterolemia (ODYSSEY COMBO II)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC11569; U1111-1121-4315 (Other: UTN); 2011-004130-34 (EudraCT Number)
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Results first posted 2015-11-06 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-06

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alirocumab 75 /up to 150 mg Q2W (Experimental): Alirocumab 75 mg every 2 weeks (Q2W) and oral placebo capsule for ezetimibe daily added to stable Lipid Modifying Therapy (LMT) for 104 weeks. Alirocumab dose up-titrated to 150 mg from Week 12 when LDL-C level ≥70 mg/dL (1.81 mmol/L) at Week 8.
  Interventions: Drug: Alirocumab; Drug: Placebo (for ezetimibe); Drug: Lipid Modifying Therapy (LMT)
- Ezetimibe 10 mg (Active Comparator): Ezetimibe 10 mg capsule daily and subcutaneous placebo for alirocumab Q2W added to stable LMT for 104 weeks.
  Interventions: Drug: Placebo (for alirocumab); Drug: Ezetimibe; Drug: Lipid Modifying Therapy (LMT)

INTERVENTIONS:
Drug: Alirocumab — 1 mL subcutaneous injection in the abdomen, thigh, or outer area of the upper arm by self-injection or by another designated person using the autoinjector.
  Other Names: REGN727/SAR236553; Praluent
  Arms: Alirocumab 75 /up to 150 mg Q2W
Drug: Placebo (for alirocumab) — 1 mL subcutaneous injection in the abdomen, thigh, or outer area of the upper arm by self-injection or by another designated person using the autoinjector.
  Arms: Ezetimibe 10 mg
Drug: Ezetimibe — One over-encapsulated tablet orally once daily at approximately the same time of the day with or without food.
  Arms: Ezetimibe 10 mg
Drug: Placebo (for ezetimibe) — One capsule once daily orally at approximately the same time of the day with or without food.
  Arms: Alirocumab 75 /up to 150 mg Q2W
Drug: Lipid Modifying Therapy (LMT) — Statin (rosuvastatin, simvastatin or atorvastatin) at stable dose.

SUMMARY:
Alirocumab (SAR236553/REGN727) is a fully human monoclonal antibody that binds PCSK9 (proprotein convertase subtilisin/kexin type 9).

Primary Objective of the study:

To demonstrate the reduction of low-density lipoprotein cholesterol (LDL-C) by alirocumab as add-on therapy to stable maximally tolerated daily statin therapy in comparison with ezetimibe after 24 weeks of treatment in participants with hypercholesterolemia at high cardiovascular (CV) risk.

Secondary Objectives:

* To evaluate the effect of alirocumab in comparison with ezetimibe on LDL-C at other time points
* To evaluate the effect of alirocumab on other lipid parameters
* To evaluate the safety and tolerability of alirocumab

DETAILED DESCRIPTION:
The maximum study duration was 115 weeks per participant, including a 3-week screening period, 104-week randomized treatment period and 8-week follow-up period.

ELIGIBILITY:
Inclusion criteria:

Participants with hypercholesterolemia and established coronary heart disease (CHD) or CHD risk equivalents who were not adequately controlled with a maximally tolerated daily dose of statin at stable dose for at least 4 weeks prior to the screening visit (Week -2).

Exclusion criteria:

* Age < 18 or legal age of adulthood, whichever was greater
* Participants without established CHD or CHD risk equivalents
* LDL-C <70 mg/dL (<1.81 mmol/L) and participants with a history of documented cardiovascular disease
* LDL-C <100 mg/dL (<2.59 mmol/L) and participants without a history of documented CV disease
* Fasting serum triglycerides >400 mg/dL (>4.52 mmol/L)

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2012-08; Primary Completion 2014-05 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (126):
- United States (58):
  - Investigational Site Number 840980, Birmingham, Alabama
  - Investigational Site Number 840918, Phoenix, Arizona
  - Investigational Site Number 840925, Tucson, Arizona
  - Investigational Site Number 840959, Anaheim, California
  - Investigational Site Number 840301, Beverly Hills, California
  - Investigational Site Number 840933, Chino, California
  - Investigational Site Number 840991, Lincoln, California
  - Investigational Site Number 840979, Los Angeles, California
  - Investigational Site Number 840952, Palm Springs, California
  - Investigational Site Number 840930, Thousand Oaks, California
  - Investigational Site Number 840921, Vista, California
  - Investigational Site Number 840962, Boynton Beach, Florida
  - Investigational Site Number 840987, Bradenton, Florida
  - Investigational Site Number 840302, Clearwater, Florida
  - Investigational Site Number 840935, Jacksonville, Florida
  - Investigational Site Number 840903, Miami, Florida
  - Investigational Site Number 840920, Miami, Florida
  - Investigational Site Number 840943, Ocala, Florida
  - Investigational Site Number 840981, Oveido, Florida
  - Investigational Site Number 840961, Port Orange, Florida
  - Investigational Site Number 840303, Sarasota, Florida
  - Investigational Site Number 840986, St. Petersburg, Florida
  - Investigational Site Number 840988, St. Petersburg, Florida
  - Investigational Site Number 840995, Meridian, Idaho
  - Investigational Site Number 840902, Evansville, Indiana
  - Investigational Site Number 840960, Topeka, Kansas
  - Investigational Site Number 840940, Oxon Hill, Maryland
  - Investigational Site Number 840966, Fall River, Massachusetts
  - Investigational Site Number 840917, Kansas City, Missouri
  - Investigational Site Number 840998, St Louis, Missouri
  - Investigational Site Number 840946, Butte, Montana
  - Investigational Site Number 840914, Lincoln, Nebraska
  - Investigational Site Number 840949, Albuquerque, New Mexico
  - Investigational Site Number 840974, New Windsor, New York
  - Investigational Site Number 840955, Greenville, North Carolina
  - Investigational Site Number 840938, Lexington, North Carolina
  - Investigational Site Number 840976, Smithfield, North Carolina
  - Investigational Site Number 840985, Winston-Salem, North Carolina
  - Investigational Site Number 840963, Cincinnati, Ohio
  - Investigational Site Number 840970, Lyndhust, Ohio
  - Investigational Site Number 840906, Marion, Ohio
  - Investigational Site Number 840997, Marion, Ohio
  - Investigational Site Number 840964, Perrysburg, Ohio
  - Investigational Site Number 840913, Charleston, South Carolina
  - Investigational Site Number 840912, Greer, South Carolina
  - Investigational Site Number 840992, Summerville, South Carolina
  - Investigational Site Number 840932, Bristol, Tennessee
  - Investigational Site Number 840944, Nashville, Tennessee
  - Investigational Site Number 840994, Fort Worth, Texas
  - Investigational Site Number 840973, Houston, Texas
  - Investigational Site Number 840939, Houston, Texas
  - Investigational Site Number 840945, Sugar Land, Texas
  - Investigational Site Number 840971, Tomball, Texas
  - Investigational Site Number 840982, Orem, Utah
  - Investigational Site Number 840931, Norfolk, Virginia
  - Investigational Site Number 840984, Richmond, Virginia
  - Investigational Site Number 840928, Renton, Washington
  - Investigational Site Number 840990, Spokane, Washington
- Canada (4):
  - Investigational Site Number 124902, Brampton
  - Investigational Site Number 124914, Mirabel
  - Investigational Site Number 124903, Montreal
  - Investigational Site Number 124918, Toronto
- Denmark (9):
  - Investigational Site Number 208913, Esbjerg
  - Investigational Site Number 208914, Glostrup Municipality
  - Investigational Site Number 208905, Hellerup
  - Investigational Site Number 208911, Herlev
  - Investigational Site Number 208907, Hvidovre
  - Investigational Site Number 208901, København S
  - Investigational Site Number 208906, Køge
  - Investigational Site Number 208908, Roskilde
  - Investigational Site Number 208903, Silkeborg
- France (4):
  - Investigational Site Number 250906, Dijon
  - Investigational Site Number 250907, Montpellier
  - Investigational Site Number 250903, Nantes
  - Investigational Site Number 250905, Nîmes
- Hungary (5):
  - Investigational Site Number 348908, Budapest
  - Investigational Site Number 348901, Budapest
  - Investigational Site Number 348903, Budapest
  - Investigational Site Number 348905, Debrecen
  - Investigational Site Number 348906, Székesfehérvár
- Israel (7):
  - Investigational Site Number 376908, Holon
  - Investigational Site Number 376903, Kfar Saba
  - Investigational Site Number 376906, Ofakim
  - Investigational Site Number 376902, Petah Tikva
  - Investigational Site Number 376904, Rehovot
  - Investigational Site Number 376907, Safed
  - Investigational Site Number 376901, Tel Aviv
- Russia (15):
  - Investigational Site Number 643906, Barnaul
  - Investigational Site Number 643903, Kemerovo
  - Investigational Site Number 643927, Moscow
  - Investigational Site Number 643928, Moscow
  - Investigational Site Number 643931, Moscow
  - Investigational Site Number 643924, Moscow
  - Investigational Site Number 643932, Moscow
  - Investigational Site Number 643908, Moscow
  - Investigational Site Number 643904, Moscow
  - Investigational Site Number 643911, Orenburg
  - Investigational Site Number 643921, Ryazan
  - Investigational Site Number 643925, Saint Petersburg
  - Investigational Site Number 643922, Saint Petersburg
  - Investigational Site Number 643914, Saint Petersburg
  - Investigational Site Number 643929, Saratov
- South Africa (8):
  - Investigational Site Number 710917, Alberton
  - Investigational Site Number 710909, Bloemfontein
  - Investigational Site Number 710914, Bloemfontein
  - Investigational Site Number 710905, Cape Town
  - Investigational Site Number 710904, Cape Town
  - Investigational Site Number 710918, Middelburg
  - Investigational Site Number 710913, Pretoria
  - Investigational Site Number 710915, Somerset West
- South Korea (14):
  - Investigational Site Number 410908, Anyang-si
  - Investigational Site Number 410920, Busan
  - Investigational Site Number 410926, Daegu
  - Investigational Site Number 410923, Gwangju
  - Investigational Site Number 410909, Seoul
  - Investigational Site Number 410922, Seoul
  - Investigational Site Number 410921, Seoul
  - Investigational Site Number 410905, Seoul
  - Investigational Site Number 410901, Seoul
  - Investigational Site Number 410914, Seoul
  - Investigational Site Number 410924, Seoul
  - Investigational Site Number 410915, Suwon
  - Investigational Site Number 410913, Uijeongbu-si
  - Investigational Site Number 410927, Wŏnju
- Ukraine (2):
  - Investigational Site Number 804905, Kiev
  - Investigational Site Number 804902, Uzhhorod

REFERENCES:
- [Background] Colhoun HM, Robinson JG, Farnier M, Cariou B, Blom D, Kereiakes DJ, Lorenzato C, Pordy R, Chaudhari U. Efficacy and safety of alirocumab, a fully human PCSK9 monoclonal antibody, in high cardiovascular risk patients with poorly controlled hypercholesterolemia on maximally tolerated doses of statins: rationale and design of the ODYSSEY COMBO I and II trials. BMC Cardiovasc Disord. 2014 Sep 20;14:121. doi: 10.1186/1471-2261-14-121. PMID 25240705
- [Result] Cannon CP, Cariou B, Blom D, McKenney JM, Lorenzato C, Pordy R, Chaudhari U, Colhoun HM; ODYSSEY COMBO II Investigators. Efficacy and safety of alirocumab in high cardiovascular risk patients with inadequately controlled hypercholesterolaemia on maximally tolerated doses of statins: the ODYSSEY COMBO II randomized controlled trial. Eur Heart J. 2015 May 14;36(19):1186-94. doi: 10.1093/eurheartj/ehv028. Epub 2015 Feb 16. PMID 25687353
- [Derived] Mahmood T, Minnier J, Ito MK, Li QH, Koren A, Kam IW, Fazio S, Shapiro MD. Discordant responses of plasma low-density lipoprotein cholesterol and lipoprotein(a) to alirocumab: A pooled analysis from 10 ODYSSEY Phase 3 studies. Eur J Prev Cardiol. 2021 Jul 23;28(8):816-822. doi: 10.1177/2047487320915803. Epub 2020 Apr 10. PMID 34298554
- [Derived] Leiter LA, Tinahones FJ, Karalis DG, Bujas-Bobanovic M, Letierce A, Mandel J, Samuel R, Jones PH. Alirocumab safety in people with and without diabetes mellitus: pooled data from 14 ODYSSEY trials. Diabet Med. 2018 Dec;35(12):1742-1751. doi: 10.1111/dme.13817. Epub 2018 Oct 9. PMID 30183102
- [Derived] Ray KK, Ginsberg HN, Davidson MH, Pordy R, Bessac L, Minini P, Eckel RH, Cannon CP. Reductions in Atherogenic Lipids and Major Cardiovascular Events: A Pooled Analysis of 10 ODYSSEY Trials Comparing Alirocumab With Control. Circulation. 2016 Dec 13;134(24):1931-1943. doi: 10.1161/CIRCULATIONAHA.116.024604. Epub 2016 Oct 24. PMID 27777279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 126 centers in 10 countries. Overall, 1112 participants were screened between August 2012 and May 2013, 392 of whom were screen failures. Screen failures were mainly due to exclusion criteria met.
Pre-assignment Details: Randomization was stratified according to prior history of myocardial infarction or ischemic stroke, intensity of statin treatment and geographical region. Assignment to arms was done centrally using Interactive Voice/Web Response System in 2:1 ratio (alirocumab: ezetimibe) after confirmation of selection criteria. 720 participants were randomized.
Groups:
- Alirocumab 75 /up to 150 mg Q2W: Subcutaneous injection of alirocumab 75 mg every 2 weeks (Q2W) and oral placebo capsule for ezetimibe daily added to stable Lipid- Modifying Therapy (LMT) for 104 weeks. Alirocumab dose up-titrated to 150 mg from Week 12 when low density lipoprotein cholesterol (LDL-C) level ≥70 mg/dL (1.81 mmol/L) at Week 8.
- Ezetimibe 10 mg: Oral ezetimibe 10 mg capsule daily and subcutaneous placebo injection for alirocumab Q2W added to stable LMT for 104 weeks.
Period: Overall Study
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Started | 479 (Randomized) | 241 (Randomized)
Treated | 479 | 241
Completed | 357 | 166
Not Completed | 122 | 75
Not completed — Adverse Event | 44 | 20
Not completed — Poor compliance to protocol | 26 | 14
Not completed — Physician Decision | 1 | 3
Not completed — Participant moved | 7 | 2
Not completed — Related to auto-injector administration | 2 | 2
Not completed — Consent withdrawn by participant | 14 | 7
Not completed — Selection criteria finally not met | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 4 | 3
Not completed — Last visit outside protocol visit window | 14 | 16
Not completed — Site closure | 1 | 1
Not completed — Other than specified above | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Alirocumab 75 /up to 150 mg Q2W: Subcutaneous injection of alirocumab 75 mg Q2W and oral placebo capsule for ezetimibe daily added to stable LMT for 104 weeks. Alirocumab dose up-titrated to 150 mg from Week 12 when LDL-C level ≥70 mg/dL (1.81 mmol/L) at Week 8.
- Total: Total of all reporting groups
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg | Total
Number analyzed (Participants) | 479 | 241 | 720
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (9.4) | 61.3 (9.2) | 61.6 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 71 | 190
  Male | 360 | 170 | 530
Calculated LDL-C in mg/dL [Mean (Standard Deviation); unit: mg/dL] — Calculated LDL-C in mg/dL from Friedewald formula (LDL cholesterol = Total cholesterol - HDL cholesterol - [Triglyceride/5]).
  mg/dL | 108.6 (36.5) | 104.6 (34.1) | 107.3 (35.7)
Calculated LDL-C in mmol/L [Mean (Standard Deviation); unit: mmol/L] | 2.812 (0.945) | 2.710 (0.884) | 2.778 (0.926)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - Intent-to-treat (ITT) Analysis
Description: Adjusted Least-squares (LS) means and standard errors at Week 24 were obtained from a mixed-effect model with repeated measures (MMRM) to account for missing data. All available post-baseline data from week 4 to week 52 regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 52
Population: ITT population: all randomized participants with one baseline and at least one post-baseline calculated LDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 467 | 240
percent change | -50.6 (1.4) | -20.7 (1.9)
Statistical Analysis 1: Comparison: Alirocumab 75 /up to 150 mg Q2W vs Ezetimibe 10 mg; Alirocumab group was compared to ezetimibe group using an appropriate contrast statement; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤0.05; LS Mean Difference = -29.8, 95% CI 2-sided [-34.4 to -25.3] — Alirocumab vs. ezetimibe

2. Secondary Outcome: Percent Change From Baseline in Calculated LDL--C at Week 24 - On--Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection or 3 days after the last capsule, whichever came first).
Time Frame: From Baseline to Week 52
Population: Modified ITT population (mITT): all randomized and treated participants with one baseline and at least one post-baseline calculated LDL-C value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 464 | 235
percent change | -52.4 (1.3) | -21.8 (1.8)
Statistical Analysis 1: Comparison: Alirocumab 75 /up to 150 mg Q2W vs Ezetimibe 10 mg; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.05 level; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤0.05; LS Mean Difference = -30.6, 95% CI 2-sided [-34.9 to -26.2] — Alirocumab vs. ezetimibe

3. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from a MMRM including all available post-baseline data from week 4 to week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 467 | 240
percent change | -51.2 (1.3) | -21.8 (1.8)
Statistical Analysis 1: Comparison: Alirocumab 75 /up to 150 mg Q2W vs Ezetimibe 10 mg; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤0.05; LS Mean Difference = -29.4, 95% CI 2-sided [-33.7 to -25.1] — Alirocumab vs. ezetimibe

4. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection or 3 days after the last capsule, whichever came first).
Time Frame: From Baseline to Week 52
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 464 | 235
percent change | -52.4 (1.2) | -22.7 (1.7)
Statistical Analysis 1: Comparison: Alirocumab 75 /up to 150 mg Q2W vs Ezetimibe 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -29.7, 95% CI 2-sided [-33.8 to -25.6] — Alirocumab vs. ezetimibe

5. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo-B) at Week 24 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline Apo-B value on-or off-treatment (Apo-B ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 452 | 228
percent change | -40.7 (1.1) | -18.3 (1.5)
Statistical Analysis 1: Comparison: Alirocumab 75 /up to 150 mg Q2W vs Ezetimibe 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -22.4, 95% CI 2-sided [-26 to -18.8] — Alirocumab vs. ezetimibe

6. Secondary Outcome: Percent Change From Baseline in Apo B at Week 24 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection or 3 days after the last capsule, whichever came first).
Time Frame: From Baseline to Week 52
Population: Participants of the mITT population with one baseline and at least one post-baseline Apo B value on-treatment (Apo-B mITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 442 | 221
percent change | -42.1 (1) | -19.1 (1.4)
Statistical Analysis 1: Comparison: Alirocumab 75 /up to 150 mg Q2W vs Ezetimibe 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -23, 95% CI 2-sided [-26.5 to -19.6] — Alirocumab vs. ezetimibe

7. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline non-HDL-C value on- or off-treatment (non-HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 467 | 240
percent change | -42.1 (1.2) | -19.2 (1.7)
Statistical Analysis 1: Comparison: Alirocumab 75 /up to 150 mg Q2W vs Ezetimibe 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -22.9, 95% CI 2-sided [-26.9 to -18.9] — Alirocumab vs. ezetimibe

8. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 24 - On-Treatment Analysis
Description: as for outcome 6
Time Frame: From Baseline up to Week 52
Population: Participants of the mITT population with one baseline and at least one post-baseline non-HDL-C value on-treatment (non-HDL-C mITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 464 | 235
percent change | -43.7 (1.1) | -20.2 (1.6)
Statistical Analysis 1: Comparison: Alirocumab 75 /up to 150 mg Q2W vs Ezetimibe 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -23.5, 95% CI 2-sided [-27.2 to -19.7] — Alirocumab vs. ezetimibe

9. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Total-C) at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline Total-C value on- or off-treatment (Total-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 467 | 240
percent change | -29.3 (0.9) | -14.6 (1.2)
Statistical Analysis 1: Comparison: Alirocumab 75 /up to 150 mg Q2W vs Ezetimibe 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -14.7, 95% CI 2-sided [-17.7 to -11.7] — Alirocumab vs. ezetimibe

10. Secondary Outcome: Percent Change From Baseline in Apo-B at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: Apo-B ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 452 | 228
percent change | -39.7 (1) | -17.2 (1.3)
Statistical Analysis 1: Comparison: Alirocumab 75 /up to 150 mg Q2W vs Ezetimibe 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -22.5, 95% CI 2-sided [-25.7 to -19.2] — Alirocumab vs. ezetimibe

11. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12 - ITT Analysis
Description: as for outcome 10
Time Frame: From Baseline to Week 52
Population: Non-HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 467 | 240
percent change | -42.6 (1.1) | -20.6 (1.5)
Statistical Analysis 1: Comparison: Alirocumab 75 /up to 150 mg Q2W vs Ezetimibe 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -22, 95% CI 2-sided [-25.6 to -18.3] — Alirocumab vs. ezetimibe

12. Secondary Outcome: Percent Change From Baseline in Total-C at Week 12 - ITT Analysis
Description: as for outcome 10
Time Frame: From Baseline to Week 52
Population: Total-C ITT population
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 467 | 240
percent change | -29.4 (0.8) | -15.1 (1.1)
Statistical Analysis 1: Comparison: Alirocumab 75 /up to 150 mg Q2W vs Ezetimibe 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -14.3, 95% CI 2-sided [-17.1 to -11.6] — Alirocumab vs. ezetimibe

13. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 52 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 52 from a MMRM model including all available post-baseline data from week 4 to week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 467 | 240
percent change | -49.5 (1.5) | -18.3 (2.1)
Statistical Analysis 1: Comparison: Alirocumab 75 /up to 150 mg Q2W vs Ezetimibe 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -31.2, 95% CI 2-sided [-36.3 to -26.1] — Alirocumab vs. ezetimibe

14. Secondary Outcome: Percentage of Participants Achieving Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - ITT Analysis
Description: Adjusted percentages at Week 24 were obtained from multiple imputation approach for handling of missing data. All available post-baseline data from week 4 to week 52 regardless of status on- or off-treatment were included in the imputation model.
Time Frame: Up to Week 52
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 467 | 240
percentage of participants | 77 | 45.6
Statistical Analysis 1: Comparison: Alirocumab 75 /up to 150 mg Q2W vs Ezetimibe 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.05; Multiple imputation approach followed by Logistic regression model; Odds Ratio (OR) = 5.4, 95% CI 2-sided [3.7 to 7.9] — Alirocumab vs. ezetimibe

15. Secondary Outcome: Percentage of Participants Achieving Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - On-Treatment Analysis
Description: Adjusted percentages at Week 24 from multiple imputation approach including available post-baseline on-treatment data from week 4 to week 52 (i.e. up to 21 days after last injection or 3 days after the last capsule, whichever came first).
Time Frame: Up to Week 52
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 464 | 235
percentage of participants | 78.9 | 47.4
Statistical Analysis 1: Comparison: Alirocumab 75 /up to 150 mg Q2W vs Ezetimibe 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.05; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 5.9, 95% CI 2-sided [3.9 to 8.8] — Alirocumab vs. ezetimibe

16. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 were obtained from multiple imputation approach followed by robust regression model for handling of missing data. All available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment were included in the imputation model.
Time Frame: From baseline to Week 52
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 467 | 240
percent change | -27.8 (1.4) | -6.1 (2)
Statistical Analysis 1: Comparison: Alirocumab 75 /up to 150 mg Q2W vs Ezetimibe 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.05; Multiple imputation approach followed by robust regression model; Adjusted Mean Difference = -21.7, 95% CI 2-sided [-26.4 to -17] — Alirocumab vs. ezetimibe

17. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline HDL-C value on- or off-treatment (HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 467 | 240
percent change | 8.6 (0.8) | 0.5 (1.1)
Statistical Analysis 1: Comparison: Alirocumab 75 /up to 150 mg Q2W vs Ezetimibe 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = 8.1, 95% CI 2-sided [5.4 to 10.7] — Alirocumab vs. ezetimibe

18. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 from multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 467 | 240
percent change | -13 (1.5) | -12.8 (2)
Statistical Analysis 1: Comparison: Alirocumab 75 /up to 150 mg Q2W vs Ezetimibe 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.9117, Regression, Robust — Threshold for significance ≤ 0.05; Multiple imputation approach followed by robust regression; Adjusted Mean Difference = -0.3, 95% CI 2-sided [-5.1 to 4.6] — Alirocumab vs. ezetimibe

19. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-1 (Apo A-1) at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline Apo A-1 value on- or off-treatment (Apo A-1 ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 452 | 228
percent change | 5 (0.6) | -1.3 (0.8)

20. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 12 - ITT Analysis
Description: Adjusted means and standard errors at Week 12 from multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 467 | 240
percent change | -22.1 (1.2) | 1.1 (1.7)

21. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 12 - ITT Analysis
Description: as for outcome 10
Time Frame: From Baseline to Week 52
Population: HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 467 | 240
percent change | 8.7 (0.7) | 2.8 (1)

22. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 12 - ITT Analysis
Description: as for outcome 20
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 467 | 240
percent change | -13 (1.5) | -12.8 (2.0)

23. Secondary Outcome: Percent Change From Baseline in Apo A-1 at Week 12 - ITT Analysis
Description: as for outcome 10
Time Frame: From Baseline to Week 52
Population: Apo A-1 ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 467 | 240
percent change | 1.5 (0.5) | -2.9 (0.7)

24. Other Pre Specified Outcome: Percent Change From Baseline in Calculated LDL-C at Week 52 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 52 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection or 3 days after the last capsule, whichever came first).
Time Frame: From Baseline to Week 52
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 464 | 235
Percent change | -51.8 (1.5) | -19.7 (2.1)

25. Other Pre Specified Outcome: Percent Change From Baseline in Calculated LDL-C at Week 104 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 104 from MMRM including all available post-baseline data from Week 4 to Week 104 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 104
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 467 | 240
Percent change | -44.2 (1.7) | -15.2 (2.4)

26. Other Pre Specified Outcome: Percent Change From Baseline in Calculated LDL-C at Week 104 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 104 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 104 (i.e. up to 21 days after last injection or 3 days after the last capsule, whichever came first).
Time Frame: From Baseline to Week 104
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 /up to 150 mg Q2W | Ezetimibe 10 mg
Number analyzed (Participants) | 464 | 235
Percent change | -48.9 (1.7) | -17.0 (2.4)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to final visit (Week 112) in the study regardless of seriousness or relationship to study drugs.
Description: Reported AEs are treatment emergent that is AEs that developed/worsened during 'the treatment emergent period' (from the first dose of double-blind study drug administration [capsule or injection, whichever came first] up the day of the last double blind injection + 70 days).
Groups:
- Alirocumab 75/Up to 150 mg Q2W: Participants exposed to Alirocumab 75 /up to 150 mg Q2W added to stable LMT (mean exposition of 90 weeks).
- Ezetimibe 10 mg: Participants exposed to Ezetimibe 10 mg added to stable LMT (mean exposition of 90 weeks).
Arm/Group | Alirocumab 75/Up to 150 mg Q2W | Ezetimibe 10 mg
Serious Adverse Events (participants affected / at risk) | 124/479 | 60/241
Other Adverse Events (participants affected / at risk) | 185/479 | 90/241
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alirocumab 75/Up to 150 mg Q2W (N=479) | Ezetimibe 10 mg (N=241)
Bronchitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 9 | 1
Diverticulitis (Infections and infestations) | 3 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0
Colonic abscess (Infections and infestations) | 1 | 0
Hepatitis E (Infections and infestations) | 1 | 0
Osteomyelitis chronic (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Scrotal abscess (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Myringitis bullous (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oestrogen receptor positive breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer stage IIIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 3 | 1
Syncope (Nervous system disorders) | 2 | 4
Transient ischaemic attack (Nervous system disorders) | 3 | 0
Carotid artery stenosis (Nervous system disorders) | 2 | 0
Presyncope (Nervous system disorders) | 1 | 0
Brain injury (Nervous system disorders) | 1 | 0
Cerebrosclerosis (Nervous system disorders) | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Facial paresis (Nervous system disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Myelitis transverse (Nervous system disorders) | 1 | 0
Sensory disturbance (Nervous system disorders) | 1 | 0
Carotid artery disease (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Transient global amnesia (Nervous system disorders) | 0 | 1
Cataract (Eye disorders) | 2 | 0
Vision blurred (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
Ophthalmoplegia (Eye disorders) | 1 | 0
Cataract nuclear (Eye disorders) | 0 | 1
Cupulolithiasis (Ear and labyrinth disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 10 | 6
Acute myocardial infarction (Cardiac disorders) | 12 | 3
Atrial fibrillation (Cardiac disorders) | 4 | 2
Angina unstable (Cardiac disorders) | 9 | 6
Cardiac failure congestive (Cardiac disorders) | 4 | 0
Cardiac arrest (Cardiac disorders) | 4 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 2 | 2
Myocardial infarction (Cardiac disorders) | 3 | 0
Ventricular tachycardia (Cardiac disorders) | 2 | 1
Atrial flutter (Cardiac disorders) | 2 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 2 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Silent myocardial infarction (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Defect conduction intraventricular (Cardiac disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 2
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Aortic dissection (Vascular disorders) | 1 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 3 | 0
Abdominal hernia (Gastrointestinal disorders) | 2 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal instability (Musculoskeletal and connective tissue disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 2
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 6 | 2
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 2 | 0
Implant site haematoma (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 1 | 1
Sudden death (General disorders) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
Bacterial test positive (Investigations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alirocumab 75/Up to 150 mg Q2W (N=479) | Ezetimibe 10 mg (N=241)
Upper respiratory tract infection (Infections and infestations) | 42 | 17
Nasopharyngitis (Infections and infestations) | 23 | 15
Influenza (Infections and infestations) | 22 | 16
Dizziness (Nervous system disorders) | 28 | 18
Headache (Nervous system disorders) | 29 | 13
Hypertension (Vascular disorders) | 31 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 25 | 13
Accidental overdose (Injury, poisoning and procedural complications) | 47 | 19

LIMITATIONS AND CAVEATS:
Manual reclassification was done by the Sponsor for the "other reasons" of non-completion of study as specified in the electronic case report form (eCRF).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.